CLINICAL TRIAL: NCT02847455
Title: Efficacy and Safety of Ilaprazole for Acute Duodenal Ulcer: A Randomized,Double-Blind,Rabeprazole-Controlled,Multicenterand Phase3 Trial in China in China
Brief Title: Ilaprazole for the Treatment of Duodenal Ulcer in Chinese Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIVZON-IY-DU-0808.0
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Duodenal Ulcer
Keywords: Ilaprazole; Proton pump inhibitor; Duodenal ulcer; Acid suppression; Randomized trial
MeSH Terms: conditions — Duodenal Ulcer | interventions — ilaprazole; Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 5 mg ilaprazole (Experimental)
  Interventions: Drug: 5 mg ilaprazole
- 10 mg ilaprazole (Experimental)
  Interventions: Drug: 10 mg ilaprazole
- 10mg Rabeprazole (Active Comparator)
  Interventions: Drug: 10 mg Rabeprazole

INTERVENTIONS:
Drug: 5 mg ilaprazole — One 5-mg ilaprazole tablet (Livzon Pharm Group Inc., China) together with three placebo tablets and one placebo capsule in a package being taken orally each
  Arms: 5 mg ilaprazole
Drug: 10 mg ilaprazole — Two 5-mg ilaprazole tablets (Livzon Pharm Group Inc., China) together with two placebo tablets and one placebo capsule in a package being taken orally each morning on an empty stomach for 4 weeks
  Arms: 10 mg ilaprazole
Drug: 10 mg Rabeprazole — one 10-mg Rabeprazole tablets together with one placebo capsule in a package being taken orally each morning on an empty stomach for 4 weeks
  Arms: 10mg Rabeprazole

SUMMARY:
Patients with endoscopically diagnosed active duodenal ulcer disease were enrolled in a randomized, double-blind, parallel and dose-ranging trial. They were randomly assigned into three groups to be treated for up to four weeks and be seen at week 1, 2 and 4: three of ilaprazole, 5, 10 mg/day, and one of Rabeprazole 10 mg/day as positive control. The primary endpoint was the ulcer healing rate at week 4. Healing of ulcer was determined by its resolution from active to scarring stage. Symptoms relief was evaluated as secondary end points by using a graded score. Safety and tolerability were evaluated on basis of clinical assessments.

DETAILED DESCRIPTION:
The primary endpoint was the healing rate of ulcers, which based on post-treatment (week 4) endoscopic changes in stage of the ulcer relative to baseline (week 0) levels. Stages of the ulcers were endoscopically assessed according to the degree of ulceration, regenerating epithelialization, and scarring, which was defined as follows: A stage (active stage, A1 & A2) where A1 stage is more severe than A2 stage, H stage (healing stage, H1 & H2) where H2 stage is better than H1 stage, and S stage (scarring stage, S1 (red scar) & S2 (white scar)) where S stage is the best stage in the three stages and S2 stage is better than S1.Healing of ulcer is deemed successful if an ulcer in A stage resolved to S stage at the end of the treatment period, regardless of S1 or S2. When endoscopy demonstrated successful ulcer healing, study medication was discontinued. Patients returned at week 2, and if unhealed further endoscopic assessment would be done at week 4. Secondary endpoints included post-treatment resolution of related gastrointestinal symptoms such as upper abdominal pain, heartburn, acid regurgitation, nausea & vomiting, eructation, and increased flatus. These symptoms were recorded on a scale ranging from 0 to 3(0=none, 1=mild, 2=moderate, 3=severe) at baseline, week 1, 2, and 4. Resolution of symptoms were defined as "excellence", "effective", "improved", or "ineffective" relative to baseline levels, of which complete symptom relief or complete absence of the symptom without recurrence was deemed as "excellence". Safety assessments based mainly on the occurrence, frequency, and severity of adverse events, which were monitored throughout the duration of the study, and also based on comprehensive indexes, including physical examination, electrocardiography, and routine laboratory investigations, which were performed at baseline and repeated at the end of the treatment period. For all adverse events, where necessary, patients were withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* - Consenting patients were eligible for enrollment if they:

  1. were 18-65 years of age,
  2. had endoscopically diagnosed active duodenal ulcers within the previous 72 hours,
  3. the number of ulcers was at least one, but no more than two with the larger diameter 0.3-2.0cm.

Exclusion Criteria:

* - Patients were ineligible if they:

  1. had cancerous or complex ulcers, Zollinger-Ellison syndrome, esophageal erosion or ulcer, varices of esophagus or fundus of stomach, or pyloric stenosis,
  2. had a known history of gastric acid suppression operation, esophageal operation or peptic operation other than simple closure of perforation,
  3. had severe complications (e.g., pyloric obstruction, active bleeding under endoscope), severe other diseases of digestive tract such as Crohn's disease and ulcerative colitis, and severe other systemic diseases,
  4. were female patients who were breast feeding, pregnant, or intended to become pregnant during the study,
  5. had taken proton pump inhibitors within the 5 days or for more than three consecutive days within the two weeks immediately preceding start of study drug,
  6. participated in a clinical trial with an investigational drug or device within the past three months,
  7. had hypersensitivity or idiosyncratic reaction to omeprazole or any other benzimidazole,
  8. had alcoholic intemperance, drug addiction or any other improper habits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2008-08; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the healing rate of ulcers, which based on post-treatment (week 4) endoscopic changes in stage of the ulcer relative to baseline (week 0) levels. | week 4

SECONDARY OUTCOMES:
Secondary endpoints included post-treatment resolution of related gastrointestinal symptoms such as upper abdominal pain, heartburn, acid regurgitation, nausea & vomiting, eructation, and increased flatus. | week 4

REFERENCES:
- [Derived] Ni H, Shi J, Hu M, Zhou N, Yang S. Cost-effectiveness analysis of Anaprazole versus Ilaprazole for the treatment of duodenal ulcers in China. Front Pharmacol. 2024 Jun 7;15:1407435. doi: 10.3389/fphar.2024.1407435. eCollection 2024. PMID 38910891